CLINICAL TRIAL: NCT03216642
Title: The Study of Bacteriology and Pathogen Drug Sensitivity of Chronic Dacryocystitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wang Zhichong, cornea department chief, Sun Yat-sen University
Other Study IDs: 2017019
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Dacryocystitis; Bacteriology
Keywords: Dacryocystitis; Bacteriology; Microbial Sensitivity Tests
MeSH Terms: conditions — Dacryocystitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Secretions from the lacrimal punctum
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: bacterial culture and analysis — Specimens were collected with soft-tipped applicators of sterile cotton swabs after syphilis of lacrimal passages.
  Other Names: antibiotic susceptibility

SUMMARY:
An observational study was designed to research the bacteriology and pathogen drug sensitivity of chronic dacryocystitis in China and optimize antibiotic therapy.

DETAILED DESCRIPTION:
For patients diagnosed with chronic dacryocystitis，we will collect the secretions after lacrimal passage irrigation, note the characters of the secretions and send the secretions for bacteria culture, analysis and pathogen drug sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with chronic dacryocystitis
2. No involvement in other drug experiment in the past 1 week

Exclusion Criteria:

1. Can not cooperate the specimen collection
2. With any other eye disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted among patients with chronic dacryocystitis attending Zhongshan Ophthalmic Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-04-17 (Estimated); Study Completion 2018-04-17 (Estimated)

PRIMARY OUTCOMES:
Bacterial agents | 2 weeks
  Specimens will be collected after irrigation of the lacrimal passage and be sent for bacterial culture and bacterial analysis.

SECONDARY OUTCOMES:
Sensitivity test | 2 weeks
  The drugs tested include Penicilin, Amikacin, Azithromycin, Cefoxitin, Levofloxacin，Ofloxacin, Cefuroxime and Tobramycin.
The colour of lacrimal sac secretion | 2 weeks
  The colour of lacrimal sac secretion will be identified by the doctor during the irrigation of the lacrimal passage.
The character of lacrimal sac secretion | 2 weeks
  The lacrimal sac secretion will be classified as mucus or pus.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided